CLINICAL TRIAL: NCT06180564
Title: Anastomotic Leak Rates in Patients Undergoing Colo-rectal Surgery With or Without Intra-operative Infra-red Thermography: Pilot Randomized Controlled Study
Brief Title: Comparison of Rates of Anastomotic Leak in Patients Undergoing Colo-rectal Surgery When Bowel Perfusion and Resection Margin is Deterimined by Intra-operative Infra-red Thermography or by Conventional Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Barun Kumar Singh, Senior resident, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COLORECTAL IRT 40
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Colo-rectal Surgery; Anastomotic Leak Large Intestine; Anastomotic Leak Rectum
Keywords: Infra-red thermography; Anastomotic leak; Colo-rectal Surgery
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: . In the test group after devascularisation of the bowel segment surgeon marked the resection line using their conventional method, then IRT was used to determine the resection line using infra- red camera in rainbow display mode. Resection line was determined by abrupt colour change (corresponds to decrease in temperature >3 degree Celsius) over the visualised bowel wall. Margins were revised if difference between surgeon and IRT determined resection lines were more than 1cm apart.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intra-operative Infra-red thermography (Experimental): . In the test group after devascularisation of the bowel segment surgeon marked the resection line using their conventional method, then IRT was used to determine the resection line using infra- red camera in rainbow display mode. Resection line was determined by abrupt colour change (corresponds to decrease in temperature >3 degree Celsius) over the visualised bowel wall. Margins were revised if difference between surgeon and IRT determined resection lines were more than 1cm apart.
  Interventions: Other: Intra-operative Infra-red thermography
- Conventional without Infra-red thermography (No Intervention): Resection margin determined by conventional visual and palpatory method

INTERVENTIONS:
Other: Intra-operative Infra-red thermography — . In the test group after devascularisation of the bowel segment surgeon marked the resection line using their conventional method, then IRT was used to determine the resection line using infra- red camera in rainbow display mode. Resection line was determined by abrupt colour change (corresponds to decrease in temperature >3 degree Celsius) over the visualised bowel wall. Margins were revised if difference between surgeon and IRT determined resection lines were more than 1cm apart.
  Arms: Intra-operative Infra-red thermography

SUMMARY:
Pilot RCT with 20 patients in both test and control group. In the control group resection & anastomosis was done using the conventional method. In the test group after devascularisation the resection line was marked on the bowel wall and IRT done using a forward looking infra- red camera with a rainbow display. Resection line was determined by a sharp change in colour on the display screen (corresponding to > 30C change in surface temperature) over the visualised bowel wall. Margins were revised if difference between surgeon and IRT determined resection lines were more than 1cm apart. Anastomosis was done as per surgeon's preference.AL was the primary outcome measure. Hospital stay, operative time, blood loss, post-operative complications as per Clavien-Dindo classification were the secondary outcome measures.

DETAILED DESCRIPTION:
A pilot randomised control study was done on adult patients undergoing elective open and lap-assisted colo-rectal surgery with ileo-colic, colo-colic, colo-rectal and colo-anal anastomoses. Patients who did not consent, who were operated in emergency, pouch surgeries and in whom resection and anastomosis was not performed were excluded.

43 patients operated between August' 2021 to November' 2022 were allocated to test and control group by simple randomisation without blinding. In the test group after mesenteric devascularisation, the site of resection was marked by the operating surgeon. After that IRT was performed using Infra-red thermal imaging FLIR C2 portable camera in the video mode and the images seen in rainbow colour display mode. The bowel segments of interest were examined from a distance range of 6 to 12 inches at the standard operation theatre temperature and humidity. Colour mapping and corresponding temperature changes were used to demarcate vascularized and non-vascularized segments of bowel. IRT-guided resection line was assigned to the place where the greatest temperature "jump" was observed (corresponding to a change of >3oC and a sharp change of colour on the screen). The IRT determined resection line was compared with the position of the resection line determined by the surgeon using conventional method. A difference of greater than 1 cm between the IRT and surgeon determined resection line was classified as non-matching and the margin was revised till the difference was less than 1 cm. The process was repeated at proximal and distal resection margins. In the control group the resection line was determined by conventional visual and palpatory method. In both the groups after resection of bowel, anastomosis was done as per surgeon preference. Diverting loop ileostomy was done on surgeon's discretion. Occurrence of an anastomotic leak (AL) up-to 8weeks post-operatively was recorded as the primary outcome. AL was defined as at-least one of the following (i) Anastomotic defect noted on physical examination. (ii) Anastomotic defect confirmed in the operating room. (iii) Anastomotic defect seen on proctoscopy. (iv) Radiologic evidence of a leak consisting of either a defect in the anastomosis and an adjacent fluid collection or stranding or extravasation of rectal contrast into the extraluminal space. (v) Clinical evidence of leak such as feculent output from abdominal/pelvic drain. Operative time, blood loss, length of hospital-stay, 30-day mortality and post-operative complications as per the Clavien-Dindo scale were the secondary outcome measured.

ELIGIBILITY:
Inclusion Criteria: Elective colo-rectal surgery, Laparoscopy assisted/ Open , Resection anastomosis done -

Exclusion Criteria: Emergency, Pouch surgery, Consent refusal, No resection & anastomosis

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2022-11-22 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Anastomotic leak | 8 weeks
  Anastomotic leak detected clinically or radiologically

SECONDARY OUTCOMES:
Clavien Dindo Complication grade | 8 weeks
  All post-operative complications
Hospital stay | 8 weeks
  From the time of surgery to discharge

OTHER OUTCOMES:
Mortality | 30 day
  Post operative mortality
Operative time and blood loss | 1 day
  From incision to closure

CONTACTS AND LOCATIONS:
Overall Officials: Barun Kumar Singh, MS, Principal Investigator — Sir Gangaram Hospital
Locations (1):
- Sir Gangaram Hospital, Delhi, India